CLINICAL TRIAL: NCT01633983
Title: Phase 2 Study of Escalating Oral Methotrexate for Central Serous Chorioretinopathy
Brief Title: Methotrexate for Central Serous Chorioretinopathy Treatment Trial
Acronym: MTX4CSC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Edward Averbukh (Other)
Responsible Party: Sponsor-Investigator, Edward Averbukh, Head of Hadassah Mt Scopus Ophthalmology Center, Hadassah Medical Organization
Organization: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: khateb-HMO-CTIL
Record Dates: First submitted 2012-07-02; First posted 2012-07-06 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Central Serous Chorioretinopathy
Keywords: Central Serous Chorioretinopathy; Methotrexate
MeSH Terms: conditions — Central Serous Chorioretinopathy | interventions — Methotrexate; Treatment Delay; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methotrexate (Experimental): Chronic CSC will be given an immediate MTX treatment
  Interventions: Drug: Methotrexate
- Delayed treatment (Experimental): Acute CSC will be followed for 3 months for a spontaneous resolution before the treatment is offered
  Interventions: Drug: Delayed treatment

INTERVENTIONS:
Drug: Methotrexate — 7.5 mg per week p.o. escalating up to 15 mg per week
  Arms: Methotrexate
Drug: Delayed treatment — Methotrexate 7.5 mg per week per os escalating to 15 mg per week
  Other Names: Methotrexate; Observation
  Arms: Delayed treatment

SUMMARY:
Central serous chorioretinopathy (CSC) is a disease of unknown origin however multiple reports have indicated correlation of appearance of CSC with exposure to exogenous or elevated levels of endogenous corticosteroid. Since the level of endogenous corticosteroids is upregulated in many inflammatory conditions, control of the inflammation may be beneficial in reducing this level thus eliminating the stimulus for CSC. Methotrexate (MTX) is widely used to control different types of inflammation. The investigators are going to try an escalating doses of MTX to treat CSC under full medical supervision.

DETAILED DESCRIPTION:
Central serous chorioretinopathy (CSC) is a disease of unknown origin usually affecting the center of the macula in adults of working age. Though previously the condition was considered stress-related, multiple recent reports have indicated correlation of appearance of CSC with exposure to exogenous or elevated levels of endogenous corticosteroid. Since the level of endogenous corticosteroids is upregulated in many inflammatory conditions, control of the inflammation may downregulate the endogenous steroids thus eliminating the stimulus for CSC. Methotrexate (MTX) is widely used to control different types of inflammation. Few short retrospective series of beneficial effect of MTX on CSC were reported recently. The investigators are going to try an escalating doses of MTX to treat CSC under full medical supervision in a prospective manner.

ELIGIBILITY:
Inclusion Criteria:

* Central Serous Chorioretinopathy

Exclusion Criteria:

* Pregnancy
* Liver disease
* Kidney disease
* Steroid use

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Optical Coherence Tomography indicating the level of central serous detachment | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Edward Averbukh, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Hebrew Univercity Medical Center, Jerusalem, Israel, Israel